CLINICAL TRIAL: NCT02170961
Title: Study of Polymorphisms of Renin Angiotensin Aldosteron Systemv(RAAS) and Matrice Metallo Protesase (MMPs) in Acute Heart Failure (AHF)
Brief Title: Study of Polymorphisms of RAAS and MMPs in Acute Heart Failure
Acronym: PRA-MMP
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Other Study IDs: PRA-MMP
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Acute Heart Failure
Keywords: Acute heart failure; RAAS; MMP3; MMP12; Polymorphysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — arterial blood samples collected in EDTA tubes and stored in - 20°C envirement for DNA extraction with salting out methods.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- acute heart failure (AHF): patients consulting the emergency department for dyspnea. the diagnosis of AHF was based on clinical, biological (BNP) and echocardiographic data.
- Non acute heart failure (NAHF): patients consulting the emergency department for dyspnea. the diagnosis of AHF was based on clinical, biological (BNP) and echocardiographic data.

SUMMARY:
this study aim to investigate the:

* association of RAAS polymorphisms and AHF
* association of MMP 3 and 12 polymorphisms and AHF

DETAILED DESCRIPTION:
Heart failure can be defined as a complex clinical syndrome that results from any structural or functional disorder of the heart, with impairment of ability to fill the ventricles or eject blood. The main event of the IC is dyspnea and fatigue, which limit exercise tolerance and induces water retention.

The renin angiotensin aldosterone system governs the salt and water homeostasis in the body. Renin is a proteolytic enzyme secreted by the juxtaglomerular apparatus of the kidney (area near the glomeruli). Renin has no direct action on the organism, but that is part of the renin-angiotensin system or the renin-angiotensin-aldosterone system is known.

To date, few published studies have examined the association between the polymorphism AGT M235T * and cardiac dysfunction; and available results are contradictory. What is not known yet is the ratio of this polymorphism with the prognosis of heart failure.

ELIGIBILITY:
Inclusion Criteria:

* aged more than 18 year old.
* acute non traumatic dyspnea .

Exclusion Criteria:

* ECG diagnostic for acute myocardial infarction or ischemic chest pain within the prior 24 hours
* a history of a heart transplant, pericardial effusion, chest wall deformity suspected of causing dyspnea
* coma, shock,MV,vasopressor drugs
* arrhythmia serious and sustained,
* pace maker
* severe mitral valve disease,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute onset dyspnea patients
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
mortality RAAS | one year
  the association between RAAS genes polymorphisms and mortality at one year average

SECONDARY OUTCOMES:
association between RAAS polymorphism and AHF | at admission (an average of 1 day)
  the association between the diagnosis of AHF (based on clinical, BNP, and echocardiographic finds) and the RAAS genes polymorphism is studied at patient admission for acute dyspnea.
association between MMP polymorphism and AHF | at admission (average of 1 day)
  the association between the diagnosis of AHF (based on clinical, BNP, and echocardiographic finds) and the MMP genes polymorphism is studied at patient admission for acute dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Samir, Professor, Principal Investigator — University of Monastir
Locations (1):
- Nouira Samir, Monastir, Emergency Department Monastir, Tunisia 5000, Tunisia

REFERENCES:
- See also: official website — http://www.urgencemonastir.com